CLINICAL TRIAL: NCT00682253
Title: Use og Bone Scintigraphy, CT and MRI for Detection of Metastases in Patients With Breast Cancer
Brief Title: Use of Bone Scintigraphy, CT and MRI in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Anni Eskild-Jensen, Aarhus University Hospital
Other Study IDs: SKF-0805
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Breast Neoplasms
Keywords: SPECT/CT; MRI; Breast neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A new imaging modality combining CT and tomographic bone scintigraphy (SPECT/CT) has enabled the combination of functional and anatomical imaging. Its use in cancer patients has not yet been evaluated or validated against a relative gold stand or clinical follow up. The purposes of this study are: 1: to validate the use of conventional planar bone scintigraphy and SPECT combined with low-dose or diagnostic CT and compare this to 3 Tesla MRI and clinical follow up. 2: to compare the specificity of low-dose and diagnostic CT, respectively, combined with bone SPECT. 3: to construct an algorithm for optimal evaluation of disease dissemination in breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histological verified breast cancer
* Age 18-80 years
* Investigation for metastases using imaging modality/modalities planned
* Written consent to participate in trial

Exclusion Criteria:

* Overweight limiting the use of MRI
* Metal parts in body
* Claustrophobia
* Allergy to contrast agents used in trial
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women aged 18-80 years with suspicision of disseminated breast cancer seen at Dept. of Oncology, Aarhus University Hospital
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark